CLINICAL TRIAL: NCT04149106
Title: Effectiveness of Seasonal Malaria Chemoprevention in Koulikoro, Mali
Brief Title: Seasonal Malaria Chemoprevention With Dihydroartemisin Piperaquin vs. Sulfadoxine-pyrimethamin+Amodiaquin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Clinical Research Center, Mali (Other)
Collaborators: Tulane University (Other); University of South Florida (Other); University of Copenhagen (Other); Deakin University (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 17-0052
Record Dates: First submitted 2019-10-01; First posted 2019-11-04 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Malaria,Falciparum
Keywords: SMC; Effectiveness; SPAQ; DHAPQ; Drug resistance
MeSH Terms: conditions — Malaria, Falciparum | interventions — fanasil, pyrimethamine drug combination; Amodiaquine

STUDY DESIGN:
Intervention Model Description: A cluster randomized design will be used.
  Year 1:
  Arm 1: SPAQ for children less than 10 years old (Standard treatment) Arm2: SPAQ will be delivery to children 3 months to less than 10 years (extension of SMC to children 5-9 years with current drug) Arm 3: DHAPQ will be delivery to children 3 months to less than 10 years
  Year 2:
  Arm 1: SPAQ will be delivery to children 3 months to less than 10 years (extension of SMC to children 5-9 years with current drug) Arm2: DHAPQ will be delivery to children 3 months to less than 10 years Arm 3: Standard of care defined as SPAQ for children less than 5 years old according the NMCP national politic for malaria control
Masking Description: Any
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard (Active Comparator): The Mali National Malaria Control program has initiated SMC for children less than 5 years since 2016 (countrywide) with SPAQ. This standard care will not change in this arm
  Interventions: Drug: Sulfadoxine pyrimethamine + Amodiaquin
- SMC with SPAQ extended to older children (Active Comparator): Within this arm, SMC with SPAQ will be extended to children 5-9 years old
  Interventions: Drug: Sulfadoxine pyrimethamine + Amodiaquin
- SMC with DHAPQ (Active Comparator): Children less than 10 years within this arm will received Dihydroartemisin piperaquin for SMC instead of SPAQ
  Interventions: Drug: Dihydroartemisinin piperaquin

INTERVENTIONS:
Drug: Sulfadoxine pyrimethamine + Amodiaquin — Monthly dose of SPAQ over three days for SMC
  Other Names: SPAQ
  Arms: SMC with SPAQ extended to older children; Standard
Drug: Dihydroartemisinin piperaquin — Monthly dose of DHAPQ for SMC
  Other Names: DHAPQ
  Arms: SMC with DHAPQ

SUMMARY:
Seasonal Malaria Chemoprevention (SMC) for children less than five years old is one the high impact interventions against malaria in sub-Saharan Africa (SSA). Since 2016, the Government of Mali and partners through the National Malaria Control Program has deployed SMC countrywide during high malaria transmission season with a total of four (4) rounds per year. Sulfadoxine-Pyrimethamine (SP) with Amodiaquine (AQ) are the drugs used for SMC. However, SP is also used for Intermittent preventative treatment (IPTp) for pregnant women while AQ has been used for decades for treatment of uncomplicated malaria.

The proposed study will examine the effect of SMC with Sulfadoxine+Amodiaquine (SP+AQ) extension to older age, the efficacy of Dihydroartemisin-Piperaquine (DHA-PQ) when used for SMC, social, cultural, economic and health systems factors associated with effective implementation of SMC. The specific aims of this study are to: 1] Assess the effect of SMC (SP+AQ) on malaria incidence and infection prevalence in different age groups across sites; 2] Study the effect of SMC (DHA-PQ) compared to SMC (SP-AQ) among children less than 10 years; 3] Determine the cost-effectiveness for each treatment regimen; ) 4] Explore factors determining effective SMC implementation including coverage of children targeted to receive treatment by community distributors, receipt of a full course of treatment, perception of medications by parents and health care providers, and sustainability; and 5) Establish a district based system to identify severe cases.

The expected outcomes of this work, upon completion of our specific aims, include 1) Recommendations to Malian health officials and other partners for improving implementation of SMC and alternative drug to SP+AQ for SMC, and 2) Guidelines for routine monitoring of SMC implementation.

DETAILED DESCRIPTION:
Study Aims The primary aim of the proposed research is to compare impact of three different treatment strategies of Seasonal malaria chemoprevention (SMC) on malaria incidence in Koulikoro health district Specific aims: Assess the effect of SMC (Sulfadoxin Pyrimethamin+Amodiaquin) on malaria incidence and infection prevalence in different age groups across sites; Study the effect of SMC with Dihydroartemesinin - Piperaquin compared to SMC with Sulfadoxin Pyrimethamin+Amodiaquin among children less than 10 years; Determine the cost-effectiveness for each treatment regimen; Explore factors determining effective SMC implementation including coverage of children targeted to receive treatment by community distributors, receipt of a full course of treatment, perception of medications by parents and health care providers, and sustainability; and Establish a district-based system to identify severe cases.

Research questions and hypotheses

Primary research question:

-Is SMC extension to children 5-9 years old with Sulfadoxin Pyrimethamin+Amodiaquin more effective on reducing malaria mortality and morbidity during the high malaria transmission season? Null hypothesis (H0): There is no benefit to SMC extension to older children with Sulfadoxin Pyrimethamin+Amodiaquin over standard SMC for children less than 5 years reducing confirmed P. falciparum case incidence, infection incidence, or community parasite prevalence during malaria transmission season

Secondary research questions:

* Could Dihydroartemesinin - Piperaquin be used as an alternative drug for SMC in case of significant resistance of P. falciparum to SP? Null hypothesis (H0): Dihydroartemesinin - Piperaquin is less effective than Sulfadoxin Pyrimethamin+Amodiaquin when used for seasonal malaria chemoprevention among children < 10 years' old
* Is extension of SMC to children < 10 years associated with a decline in the proportion of infected malaria vector, and Entomological Inoculation Rates?
* Are there difference in frequency of adverse effects to children receiving Sulfadoxin Pyrimethamin+Amodiaquin vs. children receiving Dihydroartemesinin - Piperaquin?
* What are the barriers to high and effective SMC implementation and effectiveness
* What is the cost and cost-effectiveness of SMC according to target groups and drugs used?
* What is the best delivery strategy for effective implementation and community adherence to SMC Research Activities
* Mapping and census enumeration including household geolocation of the study area will be undertaken in June 2019. The household census will be completed using house-to-house enumeration. This will be used to identify 9 candidate study villages for approximately 5,000 children aged 3 months to <10 years old. From the 9 villages, three (3) study arms will be formed (3 villages per arm). Village will be randomly allocated to sites according to geographic and environmental characteristics as well as population size.
* The census data will be used as a sampling frame for conducting the enrollment and follow-on deployment of the interventions, for cohort selection and for determining the population denominator for incidence calculated using passive case detection reported through the routine surveillance system.
* Enrollment. Before SMC, all children < 10 years old will be selected to participate. A study specific consent for will be addressed to parents of children and only children of parents who voluntarily consent will be enrolled. At enrollment, finger print, facial recognition and picture of children for whom consent was obtain will be collected and study card with picture and individual ID number will be generated for each child. Fever, Anemia and malaria infection prevalence will be collected during enrollment and infected cases will be given malaria treatment according to the Mali NMPC recommandations and free of charge.
* Sensitisation of the population to the proposed study and Community. Study investigators organized a first workshop in Koulikoro to explain the study purposes and goals. Attendees to this meeting will be the Regional and District level health authorities, Director of the 9 community health centers, Malaria focal points in Koulikoro district health center, Community leaders, Community health workers and health agents of the selected study area.
* Randomisation. From the census data, the geographical and environmental characteristics of each village, Clusters will be randomize villages to study arm considering:

  * 3 levels of population: low, medium, and high stratified and 3 regions (Northern, Central, and River).
  * The first study arm will be under standard SMC
  * The second study arm will receive SMC with standard drugs for < 10 years
  * The third study arm will receive SMC with alternative drug for < 10 years
  * SMC delivery. According the National Malaria Control Program, the first round of SMC will start in July 22nd, 2019 and a total of four monthly round will be performed. This study will follow the national calendar for SMC. During each round, teams will be deployed on each site for a week to oversee the drug distribution and monitor adherence through direct and indirect observation. A post SMC household survey will be performed to assess adherence to treatment, adverse side effects and reasons for non-compliance to SMC treatment
  * Selection and training of community health workers. For each site a list of community health workers (CHWs) and Community Health Agents (CHAs) will be established. A special on-site training will be organized for each health district before the first round of SMC. Training will be on SMC treatment, doses and coverage; electronic data capture, use of RDT, prompt administration of ACTs and referral to the Community health center of complicated malaria cases) Communities will be made aware of the new duties of their CHW/CHA before the project start.
  * Implementation science. Qualitative and quantitative research methods will be applied including observations, in-depth interviews and focus group discussions to examine all of the steps in the implementation of SMC.
  * Capture costing data. SMC drugs and delivery costs will be collected following a standardized protocol to estimate the financial and economic costs of each treatment regimen. Final cost will be compare to total expenditure for malaria treatment at community level in absence of SMC.
  * Entomological collections. During malaria transmission season, a total of three mosquito collection will be performed in each study village. Collection methods will include PSC inside houses, and HLC in and out doors. Up to 100 female anophelines per site per survey will be dissected for age grading, and tested by PCR for species identification and sporozoite ELISA.
  * Environmental context. Monthly monitoring of weather (temperature, humidity, rainfall) will be undertaken. Additionally, proximity and productivity of breeding sites will be monitored monthly. Daily weather data (temperature, humidity, rainfall) will be collected from the nearest weather station on a district level.

    3. Methodology 3.1. Study sites : Koulikoro Health District, Mali is situated in southwest Mali about 50 miles (18 km) north of Bamako and 255 miles (410 km) from the Guinea border. The district maintains 21 health zones and 71 community health posts. The current population in the district is 282,570 with approximately 4% under 1 year of age and 18% between 1 and 4 years of age. The total number of villages covered by a community health center varies from 8 to 31 villages. Kolebougou is the most populous village with 34,712 persons and Souban is the smallest with only 5,085 persons. Ongoing malaria control activities include case management (rapid diagnostic tests [RDTs] and artemisinin-based combination therapy [ACT]), IPT in pregnant women, SMC, and long-lasting insecticide treated nets (LLINs). The health centers in Koulikoro District maintain clinical and laboratory research capacity and full-time staff and clinicians for malaria screening and patient care. The site was chosen as the proposed research because of its diverse range of malaria control interventions, collaborative research agreements with USTTB, high malaria transmission rates, and rural location. All data for this project will be collected at Koulikoro Health District sites. According to geographical location, the 9 study sites are: Gouni, Kenenkou, Kamani, Doumba, Sinzani, Koula, Sirakorola, Monzombala and Chola.
  * Along the River Niger: Gouni, Kenenkou and Kamani
  * Central zone: Doumba, Koula and Sinzani
  * Northern zone: Sirakorola, Monzombala and Chola 3.2. Study Design: A cluster randomized design will be used. A total of three treatment arms will be formed (see the graphic below): Arm 1: Standard of care defined as Sulfadoxin Pyrimethamin+Amodiaquin for children less than 5 years old according the NMCP national politic for malaria control Arm2: Sulfadoxin Pyrimethamin+Amodiaquin will be delivery to children 3 months to less than 10 years (extension of SMC to children 5-9 years with current drug) Arm 3: Dihydroartemesinin - Piperaquin will be delivery to children 3 months to less than 10 years

ELIGIBILITY:
Inclusion Criteria:

* Village resident (up to the end of the malaria transmission season)
* Age 3 months to 119 month age at the time of enrollment
* Parent or guardian provided consent for their child's participant (5-14 years old)
* Absence of chronic diseases, history of allergy to SP, AQ or DHA-PQ

Exclusion Criteria:

Non resident

* Age less than 3months or greater or equal to 119 months at the time of cohort enrollment
* Presence of chronic diseases, history of allergy to SP, AQ or DHA-PQ
* Does not provide consent/assent required according to age to participate in the study

Ages: 3 Months to 119 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4556 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Malaria incidence among cohort in 2 years period | 2 years
  The incidence of malaria (uncomplicated or severe malaria): Uncomplicated malaria being defined as symptomatic malaria parasitaemia with no signs of severity and/or evidence of vital organ dysfunction measured by: (1) rapid diagnostic tests and/or (2) microscopy of blood smears. Severe malaria is defined as confirmed malaria parasitemia plus fever or history of fever (at least 37°C) plus evidence of severe/complicated pathology; e.g., convulsions, vomiting, coma, rapid (kussumal) breathing or evidence of vital organ dysfunction, and severe anemia.

SECONDARY OUTCOMES:
Malaria infection prevalence at the start and the end of malaria transmission season | 2 years
  include changes in the prevalence of P. falciparum parasitemia and anemia measured during cross-sectional surveys before SMC provision (June/July the beginning of transmission season) and after fourth round provision of SMC
Drug resistance marker prevalence in two 2 years period | 1 year
  prevalence of immunological markers for P. falciparum malaria, prevalence of molecular markers of drug resistance
SMC coverage and treatment compliance during malaria transmission season | 2 years
  total number of age eligible children sampled reporting to have received SMC and number of children who received SMC with drug metabolites in their blood divided by number of age eligible children in sample.

OTHER OUTCOMES:
Malaria control tools usage in communities | 2 years
  Estimates of the coverage and usage rates for malaria control tools (bed nets, antimalarial drugs

CONTACTS AND LOCATIONS:
Overall Officials: Seydou Doumbia, PhD, Study Director — University Clinical Research Center - USTTB - Mali
Locations (1):
- Ucrc - Usttb, Bamako, Select, Mali

IPD SHARING:
Plan to Share IPD: Yes
genomic data will be shared with Deakin University. Sharing data and resources arising from the genomics research will be a key activity of the research team. In order to prevent unnecessary duplication and to encourage collaboration, we will make the data and resources available to the malaria research community using several different means. Data arising from the research activities will be submitted to appropriate data repositories. This will include DRYAD for sample genotyping data and the GenBank for all NGS raw data. Other types of data e.g. results of sequence analyses will be published in the scientific literature. We will liaise with EuPathDB to integrate genetic, infection, and associated meta-data into EuPathDB databases. EuPathDB houses the NIH-funded Plasmodium database resource, PlasmoDB. Protocols describing new assays and laboratory methods will be published in the scientific literature. We will publish results in order to increase awareness of the scientific world.
Supporting Information: Analytic Code
Time Frame: All data and resources will be made available as soon as possible but no later than within one year of the completion of the funded project period (2021) or upon acceptance of the data for publication, or public disclosure of a submitted patent application, whichever is earlier.
Access Criteria: we will identify where the data will be available and how to access the data in any publications and presentations that we author or co-author about these data, as well as acknowledge the repository and funding source in any publications and presentations. All repositories mentioned have policies and procedures in place that will provide data access to qualified researchers or registered users, fully consistent with NIH data sharing policies and applicable laws and regulations.

REFERENCES:
- [Background] Chotsiri P, Zongo I, Milligan P, Compaore YD, Some AF, Chandramohan D, Hanpithakpong W, Nosten F, Greenwood B, Rosenthal PJ, White NJ, Ouedraogo JB, Tarning J. Optimal dosing of dihydroartemisinin-piperaquine for seasonal malaria chemoprevention in young children. Nat Commun. 2019 Jan 29;10(1):480. doi: 10.1038/s41467-019-08297-9. PMID 30696903
- [Background] Zongo I, Milligan P, Compaore YD, Some AF, Greenwood B, Tarning J, Rosenthal PJ, Sutherland C, Nosten F, Ouedraogo JB. Randomized Noninferiority Trial of Dihydroartemisinin-Piperaquine Compared with Sulfadoxine-Pyrimethamine plus Amodiaquine for Seasonal Malaria Chemoprevention in Burkina Faso. Antimicrob Agents Chemother. 2015 Aug;59(8):4387-96. doi: 10.1128/AAC.04923-14. Epub 2015 Apr 27. PMID 25918149
- [Background] Some AF, Zongo I, Compaore YD, Sakande S, Nosten F, Ouedraogo JB, Rosenthal PJ. Selection of drug resistance-mediating Plasmodium falciparum genetic polymorphisms by seasonal malaria chemoprevention in Burkina Faso. Antimicrob Agents Chemother. 2014 Jul;58(7):3660-5. doi: 10.1128/AAC.02406-14. Epub 2014 Apr 14. PMID 24733476
- [Background] Maiga H, Lasry E, Diarra M, Sagara I, Bamadio A, Traore A, Coumare S, Bahonan S, Sangare B, Dicko Y, Diallo N, Tembely A, Traore D, Niangaly H, Dao F, Haidara A, Dicko A, Doumbo OK, Djimde AA. Seasonal Malaria Chemoprevention with Sulphadoxine-Pyrimethamine and Amodiaquine Selects Pfdhfr-dhps Quintuple Mutant Genotype in Mali. PLoS One. 2016 Sep 23;11(9):e0162718. doi: 10.1371/journal.pone.0162718. eCollection 2016. PMID 27662368
- [Derived] Dicko I, Konate D, Diakite SAS, Keita B, Sanogo I, Fomba A, Traore A, Kone J, Kante S, Tessougue O, Diawara SI, Doumbia S, Diakite M. Relationship between red blood cell polymorphisms and effectiveness of seasonal malaria chemoprevention in 2020 in Dangassa, Mali. Parasitol Res. 2024 Oct 14;123(10):350. doi: 10.1007/s00436-024-08372-1. PMID 39400721
- [Derived] Toure M, Shaffer JG, Sanogo D, Keita S, Keita M, Kane F, Traore B, Dabitao D, Kone A, Doumbia CO, Keating J, Yukich J, Hansson HH, Barry AE, Diakite M, Alifrangis M, Doumbia S. Seasonal Malaria Chemoprevention Therapy in Children Up To 9 Years of Age: Protocol for a Cluster-Randomized Trial Study. JMIR Res Protoc. 2024 Jan 22;13:e51660. doi: 10.2196/51660. PMID 38252481
- [Derived] Konate D, Diawara SI, Keita B, Sogoba N, Fayical M, Guindo A, Thiam S, Traore SF, Shaffer JG, Doumbia S, Diakite M. Effectiveness and Community Acceptance of Extending Seasonal Malaria Chemoprevention to Children 5 to 14 Years of Age in Dangassa, Mali. Am J Trop Med Hyg. 2021 Nov 15;106(2):648-654. doi: 10.4269/ajtmh.21-0046. PMID 34781256